CLINICAL TRIAL: NCT06424041
Title: Fecal Microbiome Transplantation From Healthy Donors to Individuals With Fibromyalgia: A Prospective Randomized, Controlled Double-Blind Study
Brief Title: Fecal Microbiome Transplantation From Healthy Donors to Individuals With Fibromyalgia
Acronym: FM-FMT-RCT
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Amir Minerbi MD, Deputy Director, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0521-23; Weston Family Foundation (Other Grant/Funding Number: Weston Family Foundation); Israel Science Foundation (Other Grant/Funding Number: Israel Science Foundation)
Record Dates: First submitted 2024-05-09; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Fecal Microbiome Transplantation (FMT); Microbiome; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: A Double-Blinded, Randomized Placebo-Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment - FMT (Active Comparator): Participants in this arm will receive a total of 5 real FMT treatments administered weekly, followed by an additional 5 maintenance FMT treatments on a monthly basis. The first induction treatment will consist of 30 grams, with subsequent treatments comprising 15 grams each.
  Interventions: Other: Fecal Microbiome Transplantation
- Sham Treatment - FMT (Sham Comparator): Participants in this arm will receive a total of 5 sham FMT treatments administered weekly, followed by an additional 5 maintenance sham FMT treatments on a monthly basis. The first induction treatment will consist of 30 grams, with subsequent treatments comprising 15 grams each.
  Interventions: Other: Sham Fecal Microbiome Transplantation

INTERVENTIONS:
Other: Fecal Microbiome Transplantation — Healthy donor fecal microbiome transplantation, following depletion of the endogenous microbial communities using antibiotics and bowel cleansing
  Arms: Active Treatment - FMT
Other: Sham Fecal Microbiome Transplantation — Capsules containing preservative solution only, following depletion of the endogenous microbial communities using antibiotics and bowel cleansing
  Arms: Sham Treatment - FMT

SUMMARY:
This study aims to investigate if a fecal microbiome transplantation (FMT) from healthy donors can reduce symptoms of fibromyalgia, a condition causing chronic pain that is difficult to treat and diagnose. Changes in the gut bacteria of women with fibromyalgia were previously reported, which might be linked to their symptoms. In mice studies, transferring gut bacteria from individuals with fibromyalgia was shown to increase sensitivity to pain, while treatment with antibiotics and transferring bacteria from healthy individuals reversed this effect. In a small open label trial in women, improvements in pain, fatigue, and sleep problems were observed after FMT. The investigators aim to perform a larger trial following a similar path. The study aims to conduct a double-blinded, randomized, placebo-controlled trial involving 80 women diagnosed with severe fibromyalgia. Half of the participants (40) will receive the active treatment, while the other half (40) will receive a sham treatment. The allocation to either group will be randomized. Throughout the study period, both the caregivers and the participants will remain unaware of their assigned groups until the study conclusion. Participants' symptoms will be documented and their blood and stool will be tested for changes in certain metabolites. If this treatment works, it could be a significant breakthrough in managing fibromyalgia and might provide new insights into its causes.

DETAILED DESCRIPTION:
A double-blind, randomized placebo-controlled study to test the therapeutic potential of encapsulated oral fecal microbiota transplantation (FMT) from healthy donors to humans with fibromyalgia.

Fibromyalgia, a chronic and debilitating syndrome characterized by widespread pain, fatigue, sleep disturbances, and cognitive dysfunction poses a significant clinical, social, and economic burden globally, with limited targeted treatment options available. Recent studies have shed light on the potential role of the gut microbiome in fibromyalgia pathogenesis, highlighting alterations in gut microbiome composition correlated with clinical indices of the syndrome. Building upon this knowledge, the study seeks to explore the therapeutic potential of FMT, a well-established treatment increasingly investigated across various medical conditions. Preclinical investigations in mice have shown that FMT from fibromyalgia patients induces symptoms of the syndrome, while FMT from healthy controls reverses them. Encouragingly, preliminary results from an open-label pilot clinical trial involving fibromyalgia patients receiving encapsulated oral FMT from healthy donors demonstrated significant improvements in pain intensity, symptomatic burden, and quality of life measures, with favorable safety profiles. Based on these promising findings, a prospective randomized, controlled double-blind study is proposed to further evaluate the efficacy and safety of encapsulated oral FMT from healthy individuals in fibromyalgia patients. Clinical outcomes, as well as stool and serum samples, will be extensively characterized to elucidate the mechanisms underlying the effects of FMT, including its modulation of gut microbiome composition and function. The hypotheses involve expecting clinically significant improvements in pain and other symptoms of fibromyalgia following FMT, alongside corresponding alterations in gut microbiome composition and metabolomics profiles. This study aims to contribute valuable insights into the potential role of FMT as a novel therapeutic approach for fibromyalgia, addressing an unmet need in the management of this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women aged 18-75 years.
2. Diagnosis of fibromyalgia confirmed according to the 2016 diagnostic criteria by a pain physician who is a part of the study team.
3. An average reported pain of 6 or above during the preceding week.
4. Has remained symptomatic despite receiving standard care for fibromyalgia.

Exclusion Criteria:

1. Any active inflammatory condition (rheumatic, gastrointestinal or other).
2. Malignant neoplasm in the preceding 5 years.
3. Immunosuppression due to medical condition or treatment.
4. Uncontrolled psychiatric pathology.
5. Any other clinically important condition at the discretion of the investigator.
6. Known allergy to the antibiotics or laxatives used in the preparation protocol, or severe food allergy.
7. Active infection or expected antibiotic treatment in the upcoming 3 months after inclusion.
8. Pregnancy or intention to conceive.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity at week five post-transplantation | Week five post transplantation induction
  Pain intensity will be assessed using the Visual Analogue Scale (VAS), with a score of zero indicating no pain and a score of 10 representing the worst possible pain.

SECONDARY OUTCOMES:
overall symptomatic burden | Week five post transplantation induction and then on months 1, 3, 6 after last FMT
  As measured using the Fibromyalgia Impact Questionnaire (range 0-100, higher scores indicate worse symptoms)
Anxiety and depression | Week five post transplantation induction and then on months 1, 3, 6 after last FMT
  As assessed by the Hospital Anxiety and Depression Scale questionnaire (range 0-21 for each of the domains, higher scores indicate worse symptoms)
Sleep quality | Week five post transplantation induction and then on months 1, 3, 6 after last FMT
  As assessed by the Pittsburgh Sleep Quality Inventory (range 0-21, higher scores indicate worse sleep quality).
Quantitative Sensory Testing | Week five post transplantation induction and then on months 1, 3, 6 after last FMT
  Pressure, heat and cold pain thresholds (Kg/cm^2, degrees C respectively, lower thresholds indicate increased pain sensitivity)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Minerbi, MD-PhD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, North, Israel

IPD SHARING:
Plan to Share IPD: No